CLINICAL TRIAL: NCT07102927
Title: The Effects of Virtual Reality-based Training for the Treatment of Neglect Syndrome in Stroke: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1-2022-0053
Record Dates: First submitted 2025-07-24; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Stroke ( 3 Months After Onset); Cognitive Dysfunction ( MMSE < 24 ); Unilateral Neglect Syndrome
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Experimental): In the experimental group, the virtual reality-based training program for neglect syndrom (NEGTREA) was administered once a day for 30 minutes per session.
  Interventions: Device: Virtual reality-based training for the treatment of neglect syndrom in stroke
- Care Provider (Experimental): In the control group, conventional occupational therapy was administered once a day for 30 minutes per session.
  Interventions: Behavioral: Conventional occupational therapy

INTERVENTIONS:
Device: Virtual reality-based training for the treatment of neglect syndrom in stroke — An occupational therapist provided 1:1 assistance with fitting and removing the virtual reality headset (HMD), operating the software and explaining the procedures, as well as offering physical support and movement assistance when necessary to enable participants to engage in the virtual reality-based training program for neglect syndrome.
  Following measurement of each participant's interpupillary distance, the headset (HTC VIVE PRO) was adjusted and fitted while the participant was seated. The lens distance was fine-tuned using adjustment knobs to match the individual's eyes.
  The training for neglect was performed with participants seated and wearing the headset. The NEGTREA program provided a virtual environment along with visual fixation training.
  Arms: control
Behavioral: Conventional occupational therapy — An occupational therapist conducted conventional neglect therapy in a 1:1 setting for 30 minutes per session. The therapy comprised therapist-supervised, table-top tasks carefully designed to parallel the virtual reality exercises as closely as possible.
  These table-top tasks primarily focused on promoting visual scanning and sustained attention toward the neglected hemifield through practical, goal-oriented activities such as object search and manipulation. The therapist utilized a variety of tools to facilitate and optimize patient engagement in these training.
  Arms: Care Provider

SUMMARY:
This study aims to investigate the effectiveness and underlying recovery mechanisms of a virtual reality-based training program for the treatment of neglect syndrome in stroke patients in the chronic phase (more than three months after onset).

Neglect is a neurological condition characterized by a failure to attend to stimuli presented on the side contralateral to a brain lesion, despite preserved visual acuity and visual fields. Patients with neglect commonly exhibit impairments in activities of daily living, including dressing, eating, grooming, reading, and writing, and are prone to collisions with objects on the neglected side. This syndrome is widely acknowledged as a significant negative prognostic indicator for functional recovery following stroke.

Previous treatments for neglect syndrome have shown promising results. Pizzamiglio et al. reported the effectiveness of visuo-spatial scanning training, while Julkunen et al. confirmed improvement using computer-based therapy. Frascineti et al. demonstrated benefits from prism adaptation therapy, and Robertson et al. found that activating the left limbs helped reduce neglect symptoms. Additionally, Brighina et al. reported that repetitive transcranial magnetic stimulation applied to the unaffected cerebral hemisphere effectively alleviated neglect.

Recently, computer-based diagnostic tools have been developed to more accurately quantify and objectify neglect. Among them, Kim et al. developed a 3D VR program that can be applied regardless of the severity of motor impairment on the affected side. Virtual reality provides simulated, immersive environments that allow users to interact as if in real-world settings, enabling objective and quantitative assessment of neglect symptoms. In particular, visual fixation training within VR encourages spontaneous visual exploration and focused attention toward the affected side, which has been shown to be an effective strategy in reducing neglect in stroke patients.

Virtual reality-based training has been increasingly applied clinically abroad. For example, the University of California's Institute for Creative Technologies uses VR for treating PTSD in Iraq war veterans, and the VRMC in the U.S. applies it for phobia and stress treatments. In Switzerland, programs like Mind Motion Pro are used for neuroregeneration-focused rehabilitation, and Japan has developed mediVR for trunk balance training. Although research on neglect using VR is active, it generally requires active therapist involvement. Few studies have clearly demonstrated the efficacy of VR treatment specifically in stroke patients, and VR applications in rehabilitation medicine remain relatively limited compared to psychiatric fields.

In light of this background, our research team developed a virtual reality-based training program (NEGTREA) for the treatment of neglect syndrome in stroke. To evaluate its clinical feasibility, we conducted a targeted focus group interview with four out of five stroke patients with neglect who used the program. The study found that the VR-based neglect treatment was well tolerated without adverse effects and achieved high patient satisfaction, alongside improved assessment scores before and after program participation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with right cerebral hemisphere stroke confirmed by MRI or CT, with left hemiplegia, and at least three months post-stroke 2. Patients confirmed to have unilateral neglect based on the BIT score (total BIT score ≤ 196, or subtest scores BITC ≤ 129 or BITB ≤ 67) 3. Individuals with sufficient cognitive ability to participate in virtual reality training (MMSE > 18) 4. Adults aged 19 years or older

Exclusion Criteria:

* 1. Presence of Hemianopsia 2. Impaired neck movement due to orthopedic issues or other causes 3. Visual or hearing impairments that interfere with evaluation and treatment 4. Difficulty maintaining a seating posture in a chair with a backrest and armrests 5. Presence of other medical issues that may affect general cognitive decline 6. Experiencing Cybersickness symptoms such as nausea, vomiting, eye strain, disorientation, ataxia, or dizziness repeatedly, making continued training difficult and requiring discontinuation as determined by the researcher

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Behavioral Inattention Test (BIT) | up to 1 day
  The following assessment tool, developed by Wilson et al. in 1987, is designed to screen for neglect syndrome and consists of two subtests: Conventional and Behavioral. Lower scores indicate a more severe degree of neglect. It is considered a reliable tool for identifyingneglect in stroke patients and is widely used in studies assessing the validity of research related to neglect syndrome.

SECONDARY OUTCOMES:
Line Bisection | after 7 weeks of treatment
  Line Bisection provides a quik method for evaluating neglect syndrome by requiring individuals to mark the center of a series of horizontal lines using a pencil. A consistent deviation of the bisection marks toward one side is typically interpreted as an indication of neglect syndrome.
Letter Cancellation | after 7 weeks of treatment
  Letter Cancellation offers a quick method for evaluating neglect syndrome by having individuals erase specific target letters distributed across a page among various letters using a pencil. The extent and direction of the erased letters-typically showing a bias toward one side-are used to assess the severity of neglect syndrome.
  Letter Cancellation offers a quick method for evaluating neglect syndrome by having individuals erase specific target letters distributed across a page among various letters using a pencil. The extent and direction of the erased letters-typically showing a bias toward one side-are used to assess the severity of neglect syndrome.
  Letter Cancellation offers a quick method for evaluating neglect syndrome by having individuals erase specific target letters distributed across a page among various letters using a pencil. The extent and direction of the erased letters-typically showing a bias toward one side-are used to assess the severity of neglect syndrome.
Korean Catherine Bergego Scale (K-CBS) | after 7 weeks of treatment
  K-CBS, developed by Bergego et al. in 1995, is a checklist designed to evaluate the presence and severity of behavioral neglect syndrome in activities of daily living. It consists of 10 items that cover tasks such as personal hygiene, dressing, eating, and wheelchair mobility. The evaluation is conducted through direct observation by a Investigator, making it a useful tool for identifying neglect syndrome in real-life functional contexts.
MRI data(T1 weighted image, Diffusion Tensor Image, resting state functional MRI) | after 7 weeks of treatment
  This study investigate the recovery mechanisms of neglect syndrome by conducting MRI scans((T1 weighted image, Diffusion Tensor Image, resting state functional MRI) before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No